CLINICAL TRIAL: NCT03019055
Title: Phase 1/1b Study of Redirected Autologous T Cells Engineered to Contain an Anti CD19 and Anti CD20 scFv Coupled to CD3ζ and 4-1BB Signaling Domains in Patients With Relapsed and/or Refractory CD19 or CD20 Positive B Cell Malignancies
Brief Title: Study of CAR-20/19-T Cells in Patients With Relapsed Refractory B Cell
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Nirav Shah, Associate Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00028724
Record Dates: First submitted 2017-01-05; First posted 2017-01-12 (Estimated); Results first posted 2021-05-07 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: CAR-T; Chimeric antigen receptor T-cell therapy; CAR Therapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Intervention Model Description: The study is divided into two phases. Phase 1 and Phase 1b. Phase 1: consists of 2 cohorts; dose escalation and dose expansion. The CAR-T cells were given over 2 days.
  In the phase 1 portion, there will be a dose escalation cohort to determine the safe CAR-20/19-T cell dose in patients with CLL/SLL and NHL. Once the desired dose has been identified there will be a 6 patient dose expansion phase at the specified dose level.
  Phase 1b: In the Phase 1b portion of the study, we will test the safety of unfractionated CAR-T cells utilizing the safe dose identified in the phase 1 portion (2.5 x 10^6 cells/kg).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CAR-20/19-T cells (1.0 x10^5 CAR-20/19-T cells/kg) (Experimental): Dose Escalation Phase: CAR-20/19-T transduced with a lentiviral vector to express an anti CD19 and anti CD20 tandem receptor coupled to CD3ζ and 4-1BB signaling domains will be administered by IV injection. Patients will receive one of four dose levels based the study protocol. Cells will be given over 2 days, 30% of cells infused on Day 0 and 70% of cells infused on Day 1 in the Phase 1 portion and as a single infusion in the Phase 1b portion.
  Interventions: Biological: CAR-20/19-T cells (1.0 x10^5 CAR-20/19-T cells/kg)
- CAR-20/19-T cells (2.5 x10^5 CAR-20/19-T cells/kg) (Experimental): Dose Escalation Phase: CAR-20/19-T transduced with a lentiviral vector to express an anti CD19 and anti CD20 tandem receptor coupled to CD3ζ and 4-1BB signaling domains will be administered by IV injection. Patients will receive one of four dose levels based the study protocol. Cells will be given over 2 days, 30% of cells infused on Day 0 and 70% of cells infused on Day 1 in the Phase 1 portion and as a single infusion in the Phase 1b portion.
  Interventions: Biological: CAR-20/19-T cells (2.5 x10^5 CAR-20/19-T cells/kg)
- CAR-20/19-T cells (7.5 x10^5 CAR-20/19-T cells/kg) (Experimental): Dose Escalation Phase: CAR-20/19-T transduced with a lentiviral vector to express an anti CD19 and anti CD20 tandem receptor coupled to CD3ζ and 4-1BB signaling domains will be administered by IV injection. Patients will receive one of four dose levels based the study protocol. Cells will be given over 2 days, 30% of cells infused on Day 0 and 70% of cells infused on Day 1 in the Phase 1 portion and as a single infusion in the Phase 1b portion.
  Interventions: Biological: CAR-20/19-T cells (7.5 x10^5 CAR-20/19-T cells/kg)
- CAR-20/19-T cells (2.5 x10^6 CAR-20/19-T cells/kg) (Experimental): Dose Escalation Phase: CAR-20/19-T transduced with a lentiviral vector to express an anti CD19 and anti CD20 tandem receptor coupled to CD3ζ and 4-1BB signaling domains will be administered by IV injection. Patients will receive one of four dose levels based the study protocol. Cells will be given over 2 days, 30% of cells infused on Day 0 and 70% of cells infused on Day 1 in the Phase 1 portion and as a single infusion in the Phase 1b portion.
  Interventions: Biological: CAR-20/19-T cells (2.5 x10^6 CAR-20/19-T cells/kg)

INTERVENTIONS:
Biological: CAR-20/19-T cells (1.0 x10^5 CAR-20/19-T cells/kg) — CAR-20/19-T cells will be administered either fresh or thawed after cryopreservation by IV injection.
  Phase 1 Dose Level 0: 2.5 x10^5 CAR-20/19-T cells/kg (starting dose level)
  Arms: CAR-20/19-T cells (1.0 x10^5 CAR-20/19-T cells/kg)
Biological: CAR-20/19-T cells (2.5 x10^5 CAR-20/19-T cells/kg) — CAR-20/19-T cells will be administered either fresh or thawed after cryopreservation by IV injection.
  Phase 1 Dose Level 1: 7.5 x10^5 CAR-20/19-T cells/kg
  Arms: CAR-20/19-T cells (2.5 x10^5 CAR-20/19-T cells/kg)
Biological: CAR-20/19-T cells (7.5 x10^5 CAR-20/19-T cells/kg) — CAR-20/19-T cells will be administered either fresh or thawed after cryopreservation by IV injection.
  Phase 1 Dose Level 2: 2.5 x10^6 CAR-20/19-T cells/kg (goal cell dose)
  Phase 1b Expansion Dose Level: 2.5 x 10^6 cells/kg (single infusion)
  Arms: CAR-20/19-T cells (7.5 x10^5 CAR-20/19-T cells/kg)
Biological: CAR-20/19-T cells (2.5 x10^6 CAR-20/19-T cells/kg) — CAR-20/19-T cells will be administered either fresh or thawed after cryopreservation by IV injection.
  Arms: CAR-20/19-T cells (2.5 x10^6 CAR-20/19-T cells/kg)

SUMMARY:
This is a phase 1/1b, interventional single arm, open label, treatment study designed to evaluate the safety and feasibility of infusion of autologous T cells engineered to contain an anti-cluster of differentiation 19 (CD19) and anti-cluster of differentiation 20 (CD20) single chain variable fragment (scFv) coupled to cluster of differentiation CD3ζ (CD3ζ) and co-stimulatory domain 4-1BB (4-1BB) signaling domains in patients with relapsed and/or refractory CD19 or CD20 positive B cell malignancies

DETAILED DESCRIPTION:
This is a single center, single arm, open label phase I/1b study to demonstrate the feasibility of manufacturing CAR-T cells expressing tandem receptors against both CD20 and CD19 (CAR-20/19-T) in a completely closed system using the CliniMACS Prodigy device and then determine the safety of this dual targeted CAR in a first-in-human study of patients with relapsed and refractory B cell malignancies. Secondary outcomes will include response rates, and observed toxicities of the treatment, specifically the development of cytokine release syndrome (CRS), an inflammatory storm that has been seen with previous CAR-T therapies.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of B-cell non-Hodgkin lymphoma (NHL) or chronic lymphocytic leukemia (CLL) / small lymphocytic leukemia (SLL): Patients must be aged≥18 years with relapsed, refractory disease and no available curative options that meet clinical criteria to initiate treatment.
2. Patients with B-cell NHL or CLL/SLL must have either CD19 or CD20 positive disease on most recent biopsy performed (a repeat biopsy is not mandatory for this study except as noted below). A minimum of 5% CD19 or CD20 positivity by immunohistochemistry or flow cytometry on prior or repeat biopsy is required.
3. Absolute CD3+ T cell count ≥50/mm^3.
4. MRI brain and Lumbar Puncture with cerebral spinal fluid (CSF) analysis by cytology and flow cytometry without evidence of central nervous system (CNS) involvement only in patients with history of CNS involvement.
5. Measurable disease must have been documented within 4 weeks of the time of consent defined as the following by disease specific subtype:

   1. B-cell NHL: Active disease defined as nodal lesions greater than 20 mm in the long axis or extranodal lesions >10 mm in long and short axis or bone marrow involvement that is biopsy proven.
   2. CLL/SLL: Active disease by either bone marrow, peripheral flow cytometry, or CT and/or positron emission tomography (PET) imaging with nodal disease.
6. Patients should have failed at least two lines of a standard treatment and meet disease specific criteria detailed below:

   1. CLL/SLL: measurable disease as defined above that has relapsed after at least one line of chemo-immunotherapy and progressed or intolerant to ibrutinib monotherapy.
   2. CD19 or CD20 positive B cell NHL limited to the following histologies: Advanced Stage III or IV Follicular Lymphoma, Diffuse Large B cell Lymphoma and associated subtypes (e.g. aggressive B-cell lymphoma, T-cell/histocyte rich B-cell lymphoma, primary mediastinal B-cell lymphoma, Epstein Barr virus positive diffuse large B-cell lymphoma, transformed lymphoma such as transformed follicular or marginal zone lymphoma, and Richter's transformation) and Mantle cell lymphoma. Specific criteria include:

      * Patients must have active, measurable disease after two lines of cytotoxic chemotherapy of which one must be anthracycline containing.
      * Must have received Rituximab or another CD20 antibody and at minimum two chemotherapy regimens appropriate for their disease.
      * Either failed autologous transplant or ineligible to receive autologous transplant
7. Karnofsky performance score ≥70. See Appendix A for scales.
8. Normal Baseline Neurological Evaluation: Mini-Mental Status Exam Score 24-30.
9. Adequate hepatic function, defined as aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <5 x upper limit of normal (ULN); serum bilirubin and alkaline phosphatase <5 x ULN, or considered not clinically significant as per the clinical PIs discretion (e.g. Gilbert's or indirect hyperbilirubinemia) or felt to be due to underlying disease.
10. Adequate renal function, defined as creatinine clearance>60 ml/min
11. Able to provide written informed consent.
12. Agree to practice birth control during the study.
13. Adequate cardiac function as indicated by New York Heart Association (NYHA) classification I or II AND left ventricular ejection fraction of ≥35% (by echocardiogram or MUGA) and adequate pulmonary function as indicated by room air oxygen saturation of ≥92%.
14. Expected survival >12 weeks.
15. Negative urine or serum pregnancy test in females of child bearing potential at study entry and again within 48 hours' prior lymphodepleting chemotherapy.
16. Patients with prior blinatumomab treatment require repeat biopsy post-blinatumomab treatment that demonstrates CD19 or CD20 positive disease.
17. Meet criteria for regarding fertility and contraception.
18. Central line access will be required for CAR-20/19-T cell infusion.

Exclusion Criteria

1. Positive beta-human chorionic gonadotropin in females of child-bearing potential.
2. Patients with known systemic allergy to bovine or murine products.
3. Known prior positive serology for human anti-mouse antibody (HAMA).
4. Confirmed active human immunodeficiency virus (HIV), Hepatitis B or C infection.
5. History of significant autoimmune disease OR active, uncontrolled autoimmune phenomenon: such as systemic lupus erythematous, Wegner's glomerulonephritis, autoimmune hemolytic anemia, idiopathic thrombocytopenic purpura (AIHA, ITP) requiring steroid therapy defined as >20 mg of prednisone or equivalent daily.
6. Presence of ≥grade 3 non-hematologic toxicities as per CTCAE version 5.0 from any previous treatment unless it is felt to be due to underlying disease.
7. Concurrent use of investigational therapeutic agents or enrollment on another therapeutic clinical trial at any institution. Minimum of ≥4 weeks required from administration of any other investigational agents on other clinical trials prior to enrollment on this CAR-T protocol.
8. Refusal to participate in the long-term follow-up protocol.
9. Patients with active CNS involvement by malignancy on MRI or by lumbar puncture.

   a. Patients with prior CNS disease that has been effectively treated will be eligible providing treatment was >4 weeks before enrollment and a remission documented within 8 weeks of planned CAR-T cell infusion by MRI brain and CSF analysis.
10. Previous recipients of allogeneic hematopoietic stem cell transplantation (AHCT) are excluded if they are <100 days' post-transplant, have evidence of active graft-versus-host-disease (GVHD) of any grade, or are currently on immunosuppression.
11. Previous CAR-T cell therapy directed at either CD19 or CD20 within 100 days of planned CAR-20/19-T cell infusion (does not include re-enrollment)

    a. Patients with prior CAR-T treatment against CD19 or CD20 must have repeat biopsy confirming a minimum of 5% CD19 or CD20 positivity by immunohistochemistry or flow cytometry.
12. Anti-CD20 antibody treatment within 4 weeks of cell infusion.
13. Anti-CD19 antibody treatment within 4 weeks of cell infusion.
14. Cytotoxic chemotherapy other than lymphodepletion within 14 days of CAR-T cell infusion.
15. Cytotoxic chemotherapy treatment within 14 days or steroid treatment (other than replacement dose steroids) within 7 days prior to apheresis collection for CAR-T cells.
16. Patients post solid organ transplant who develop high grade lymphomas or leukemias.
17. Concurrent active malignancy other than basal or squamous cell carcinomas of the skin.

Special Criteria for regarding Fertility and Contraception

Female subjects of reproductive potential (women who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or have not undergone a sterilization procedure [hysterectomy or bilateral oophorectomy]) must have a negative serum or urine pregnancy test performed as part of eligibility criteria and again within 48 hours of initiation of lymphodepleting chemotherapy.

Due to the high-risk level of this study, while enrolled, all subjects must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization). Additionally, if participating in sexual activity that could lead to pregnancy, the study subject must agree to use reliable and double barrier methods of contraception during the follow-up period of the protocol.

Acceptable birth control includes a combination of two of the following methods:

* Condoms* (male or female) with or without a spermicidal agent.
* Diaphragm or cervical cap with spermicide
* Intrauterine device (IUD)
* Hormonal-based contraception Subjects who are not of reproductive potential (women who are premenarche or have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy tubal ligation, salpingectomy, and/or bilateral oophorectomy or men who have documented azoospermia) are eligible without requiring the use of contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirav Shah, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zurko JC, Fenske TS, Johnson BD, Bucklan D, Szabo A, Xu H, Chaney K, Hamadani M, Hari P, Shah NN. Long-term outcomes and predictors of early response, late relapse, and survival for patients treated with bispecific LV20.19 CAR T-cells. Am J Hematol. 2022 Dec;97(12):1580-1588. doi: 10.1002/ajh.26718. Epub 2022 Sep 20. PMID 36068950
- [Derived] Knight JM, Szabo A, Arapi I, Wu R, Emmrich A, Hackett E, Sauber G, Yim S, Johnson B, Hari P, Schneider D, Dropulic B, Cusatis RN, Cole SW, Hillard CJ, Shah NN. Patient-reported outcomes and neurotoxicity markers in patients treated with bispecific LV20.19 CAR T cell therapy. Commun Med (Lond). 2022 May 12;2(1):49. doi: 10.1038/s43856-022-00116-5. eCollection 2022. PMID 35603278
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Shah NN, Johnson BD, Schneider D, Zhu F, Szabo A, Keever-Taylor CA, Krueger W, Worden AA, Kadan MJ, Yim S, Cunningham A, Hamadani M, Fenske TS, Dropulic B, Orentas R, Hari P. Bispecific anti-CD20, anti-CD19 CAR T cells for relapsed B cell malignancies: a phase 1 dose escalation and expansion trial. Nat Med. 2020 Oct;26(10):1569-1575. doi: 10.1038/s41591-020-1081-3. Epub 2020 Oct 5. PMID 33020647

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 31 enrolled subjects who signed the informed consent form, 26 met all eligibility criteria.
Groups:
- CAR-20/19-T Cells (1.0 x10^5 CAR-20/19-T Cells/kg): Dose Escalation Phase: CAR-20/19-T transduced with a lentiviral vector to express an anti CD19 and anti CD20 tandem receptor coupled to CD3ζ and 4-1BB signaling domains will be administered by IV injection. Patients will receive one of four dose levels based the study protocol. Cells will be given over 2 days, 30% of cells infused on Day 0 and 70% of cells infused on Day 1 in the Phase 1 portion and as a single infusion in the Phase 1b portion.
  CAR-20/19-T cells (1.0 x10^5 CAR-20/19-T cells/kg): CAR-20/19-T cells will be administered either fresh or thawed after cryopreservation by IV injection.
  Phase 1 Dose Level 0: 2.5 x10^5 CAR-20/19-T cells/kg (starting dose level)
- CAR-20/19-T Cells (2.5 x10^5 CAR-20/19-T Cells/kg): Dose Escalation Phase: CAR-20/19-T transduced with a lentiviral vector to express an anti CD19 and anti CD20 tandem receptor coupled to CD3ζ and 4-1BB signaling domains will be administered by IV injection. Patients will receive one of four dose levels based the study protocol. Cells will be given over 2 days, 30% of cells infused on Day 0 and 70% of cells infused on Day 1 in the Phase 1 portion and as a single infusion in the Phase 1b portion.
  CAR-20/19-T cells (2.5 x10^5 CAR-20/19-T cells/kg): CAR-20/19-T cells will be administered either fresh or thawed after cryopreservation by IV injection.
  Phase 1 Dose Level 1: 7.5 x10^5 CAR-20/19-T cells/kg
- CAR-20/19-T Cells (7.5 x10^5 CAR-20/19-T Cells/kg): Dose Escalation Phase: CAR-20/19-T transduced with a lentiviral vector to express an anti CD19 and anti CD20 tandem receptor coupled to CD3ζ and 4-1BB signaling domains will be administered by IV injection. Patients will receive one of four dose levels based the study protocol. Cells will be given over 2 days, 30% of cells infused on Day 0 and 70% of cells infused on Day 1 in the Phase 1 portion and as a single infusion in the Phase 1b portion.
  CAR-20/19-T cells (7.5 x10^5 CAR-20/19-T cells/kg): CAR-20/19-T cells will be administered either fresh or thawed after cryopreservation by IV injection.
  Phase 1 Dose Level 2: 2.5 x10^6 CAR-20/19-T cells/kg (goal cell dose)
  Phase 1b Expansion Dose Level: 2.5 x 10^6 cells/kg (single infusion)
Period: Overall Study
Arm/Group | CAR-20/19-T Cells (1.0 x10^5 CAR-20/19-T Cells/kg) | CAR-20/19-T Cells (2.5 x10^5 CAR-20/19-T Cells/kg) | CAR-20/19-T Cells (7.5 x10^5 CAR-20/19-T Cells/kg) | CAR-20/19-T Cells (2.5 x10^6 CAR-20/19-T Cells/kg)
Started | 0 | 3 | 3 | 20
Completed | 0 | 3 | 3 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to a lack of dose limiting toxicities at higher dosages, no subjects were enrolled in the 1.0x10^5 cell/kg dosage level.
Groups:
- Total: Total of all reporting groups
Arm/Group | CAR-20/19-T Cells (1.0 x10^5 CAR-20/19-T Cells/kg) | CAR-20/19-T Cells (2.5 x10^5 CAR-20/19-T Cells/kg) | CAR-20/19-T Cells (7.5 x10^5 CAR-20/19-T Cells/kg) | CAR-20/19-T Cells (2.5 x10^6 CAR-20/19-T Cells/kg) | Total
Number analyzed (Participants) | 0 | 3 | 3 | 20 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 52.33 (2.31) | 55.00 (8.19) | 55.85 (14.44) | 55.35 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 0 | 3 | 4
  Male |  | 2 | 3 | 17 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0 | 0 | 0
  Not Hispanic or Latino |  | 3 | 3 | 20 | 26
  Unknown or Not Reported |  | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 | 1 | 1
  Asian |  | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0 | 0
  Black or African American |  | 0 | 0 | 2 | 2
  White |  | 2 | 3 | 16 | 21
  More than one race |  | 0 | 0 | 0 | 0
  Unknown or Not Reported |  | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 3 | 3 | 20 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events After CAR 20/19-T Cell Infusion
Description: This measure is the number of adverse events with grade 3 to 5 severity per Common Terminology Criteria for Adverse Events (ver. 4.03) occurring within the first 28 days following infusion.
Time Frame: 28 days after infusion
Population: Of the eligible subjects, CAR cell product did not reach the required cell concentration for infusion for 4 subjects in the highest dosage level. These subjects were withdrawn by the investigator. Overall, 22 subjects received the investigational product in this study. The initial concentration for the study was 2.5x10^5 cells/kg. No dose limiting toxicities were experienced at this concentration and the reduced dose of 1.0x10^5 cells/kg was not used.
Measure: Number; unit: Serious Adverse Events
Arm/Group | CAR-20/19-T Cells (1.0 x10^5 CAR-20/19-T Cells/kg) | CAR-20/19-T Cells (2.5 x10^5 CAR-20/19-T Cells/kg) | CAR-20/19-T Cells (7.5 x10^5 CAR-20/19-T Cells/kg) | CAR-20/19-T Cells (2.5 x10^6 CAR-20/19-T Cells/kg)
Number analyzed (Participants) | 0 | 3 | 3 | 16
Serious Adverse Events |  | 7 | 4 | 22

ADVERSE EVENTS:
Time Frame: 28 days
Description: No subjects were enrolled in the 1.0x10^5 cells/kg dosage group.
Arm/Group | CAR-20/19-T Cells (1.0 x10^5 CAR-20/19-T Cells/kg) | CAR-20/19-T Cells (2.5 x10^5 CAR-20/19-T Cells/kg) | CAR-20/19-T Cells (7.5 x10^5 CAR-20/19-T Cells/kg) | CAR-20/19-T Cells (2.5 x10^6 CAR-20/19-T Cells/kg)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/3 | 0/3 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/0 | 3/3 | 3/3 | 16/16
Other Adverse Events (participants affected / at risk) | 0/0 | 3/3 | 3/3 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAR-20/19-T Cells (1.0 x10^5 CAR-20/19-T Cells/kg) (N=0) | CAR-20/19-T Cells (2.5 x10^5 CAR-20/19-T Cells/kg) (N=3) | CAR-20/19-T Cells (7.5 x10^5 CAR-20/19-T Cells/kg) (N=3) | CAR-20/19-T Cells (2.5 x10^6 CAR-20/19-T Cells/kg) (N=16)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAR-20/19-T Cells (1.0 x10^5 CAR-20/19-T Cells/kg) (N=0) | CAR-20/19-T Cells (2.5 x10^5 CAR-20/19-T Cells/kg) (N=3) | CAR-20/19-T Cells (7.5 x10^5 CAR-20/19-T Cells/kg) (N=3) | CAR-20/19-T Cells (2.5 x10^6 CAR-20/19-T Cells/kg) (N=16)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (13) | 2 (12) | 14 (37)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3) | 10 (15)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (8) | 6 (9)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 11 (18)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (6) | 11 (17)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 3 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (3) | 3 (7) | 12 (20)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 1 (4) | 13 (18)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1) | 6 (7)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 7 (10)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (10)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 9 (17)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (3) | 1 (2) | 3 (6)
Creatinine increased (Investigations) | 0 (0) | 2 (7) | 0 (0) | 8 (14)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (8) | 3 (15) | 16 (49)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (12) | 3 (21) | 16 (59)
Platelet count decreased (Investigations) | 0 (0) | 2 (12) | 2 (11) | 13 (32)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 3 (9) | 3 (13) | 16 (68)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (8) | 0 (0) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (6) | 9 (14)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (7)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 3 (11) | 1 (1) | 10 (27)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (6) | 1 (6) | 13 (27)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 0 (0) | 7 (16)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (7)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (8) | 1 (2) | 9 (21)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 1 (2) | 4 (6)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (10)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1) | 8 (11)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 5 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 4 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (8) | 3 (9) | 8 (13)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (3) | 7 (15)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT03019055/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT03019055/ICF_001.pdf